CLINICAL TRIAL: NCT05470361
Title: Investigating the Effects of Stellate Ganglion Block and Superior Cervical Ganglion Block on Sleep and Recovery Using Biometric Capture Devices
Brief Title: Effects of Stellate Ganglion Block and Superior Cervical Ganglion Block on Sleep and Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Whoop Inc. (Industry); Stella MSO, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: UQueenslandSGB
Record Dates: First submitted 2022-06-07; First posted 2022-07-22 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-05

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who suffer from PTSD: The sample will be composed of 30 patients from Stella's Chicago practice: 712 N Dearborn St, Chicago, Illinois 60654
  Interventions: Procedure: stellate ganglion block (SGB)

INTERVENTIONS:
Procedure: stellate ganglion block (SGB) — The protocol for the SGB plus SCGB will be followed, wherein participants are given right-side procedures followed by left-side procedures on a different day if no initial improvement is seen. This procedure is carried out by injecting a local anesthetic into the neck to target the Stellate Ganglion and Superior Cervical Ganglion nerve bundles.

SUMMARY:
The aim of this study is to discover whether the Stellate Ganglion Block (SGB) plus the Superior Cervical Ganglion Block (SCGB) procedure is associated with improvements in heart rate variability and sleep quality as measured by the Whoop biometric capture device. It is predicted that after receiving the blocks, patients will show objectively improved measures of stress in the form of higher heart rate variability and improved sleep quality as well as improved subjective wellbeing.

DETAILED DESCRIPTION:
PTSD is meaningfully related to workforce productivity and quality of life factors, including loss of employment and decreases in general life satisfaction. Trauma leads to symptoms that diminish capacity to experience warm and loving feelings for others (emotional numbness), profound negative changes in our self-image and identity, fears that often limit enjoyment of pleasurable activities, and other life-altering challenges. Many survivors experience recurrent feelings of helplessness and horror, and may commonly experience crippling panic attacks, feelings of self-blame and shame, chronically disrupted sleep, and relationship conflict with loved ones.

Low resting Heart Rate Variability (HRV)-- the variability in the time in between heart beats--is a physiological indicator of stress and has been associated with reductions in wellbeing and increases in all-cause mortality. Higher heart rate variability is associated with better sleep quality while lower heart rate variability is associated with increased chronic inflammation. The negative effects of PTSD on sleep are well-documented, and interventions are often targeted at alleviating this damaging consequence, as insufficient sleep can perpetuate anxiety and impair day-to-day functioning, leading to an overall reduced quality of life.

The current standard of care is to offer a combination of trauma-focused psychotherapy and symptom-focused medications, typically a selective serotonin reuptake inhibitor medication. However, a promising treatment known as the Stellate Ganglion Block (SGB) plus the Superior Cervical Ganglion Block (SCGB) procedure has been shown to alleviate PTSD symptoms without any of the side-effects and barriers known to patients on conventional treatments. While this treatment shows promise, most of the research performed so far has used subjective self-report measures of sleep quality and stress. Whoop biometric capture devices offer an opportunity to objectively measure sleep quality and heart rate variability to investigate the effects of the SGB. Physiological data could reveal whether this treatment works not just to alleviate subjective stress, but to physically reduce the effects of PTSD on the body.

ELIGIBILITY:
Inclusion Criteria:

- PTSD Symptoms

Exclusion Criteria:

* none

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients who have attended the practice in Chicago, have arranged to have the SGB plus SCGB procedure to address their PTSD, and are interested in monitoring their symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 8 weeks
  The primary outcome measures for the study will be participant sleep scores (derived from time spent in each sleep stage) and Heart Rate Variability, both of which will be measured by a Whoop strap biometric capture device. Higher heartrate variability represents a better outcome (healthier nervous system). Likewise a higher sleep score represents a better and more complete recovery.

SECONDARY OUTCOMES:
Self-reported Post-Traumatic Stress Disorder symptoms | 8 weeks
  Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorder (DSM-5). Scores range from 0-80. Higher scores mean worse Post-Traumatic Stress Disorder.
Self-reported depression symptoms | 8 weeks
  Beck Depression Inventory-II. Scores from 0-63. Higher scores indicate more severe depression.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkire, M. T., Hollifield, M., Khoshsar, R., Nguyen, L., Alley, S. R., & Reist, C. (2015, October). Neuroimaging suggests that stellate ganglion block improves post-traumatic stress disorder (PTSD) through an amygdala mediated mechanism. In The Anesthesiology Annual Meeting.
- [Background] Alvaro PK, Roberts RM, Harris JK. A Systematic Review Assessing Bidirectionality between Sleep Disturbances, Anxiety, and Depression. Sleep. 2013 Jul 1;36(7):1059-1068. doi: 10.5665/sleep.2810. PMID 23814343
- [Background] Bernardy NC, Friedman MJ. Psychopharmacological strategies in the management of posttraumatic stress disorder (PTSD): what have we learned? Curr Psychiatry Rep. 2015 Apr;17(4):564. doi: 10.1007/s11920-015-0564-2. PMID 25749751
- [Background] Feeny NC, Zoellner LA, Fitzgibbons LA, Foa EB. Exploring the roles of emotional numbing, depression, and dissociation in PTSD. J Trauma Stress. 2000 Jul;13(3):489-98. doi: 10.1023/A:1007789409330. PMID 10948488
- [Background] Filipas HH, Ullman SE. Child sexual abuse, coping responses, self-blame, posttraumatic stress disorder, and adult sexual revictimization. J Interpers Violence. 2006 May;21(5):652-72. doi: 10.1177/0886260506286879. PMID 16574638
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Lipov EG, Joshi JR, Lipov S, Sanders SE, Siroko MK. Cervical sympathetic blockade in a patient with post-traumatic stress disorder: a case report. Ann Clin Psychiatry. 2008 Oct-Dec;20(4):227-8. doi: 10.1080/10401230802435518. No abstract available. PMID 19034755
- [Background] Lynch JH, Mulvaney SW, Kim EH, de Leeuw JB, Schroeder MJ, Kane SF. Effect of Stellate Ganglion Block on Specific Symptom Clusters for Treatment of Post-Traumatic Stress Disorder. Mil Med. 2016 Sep;181(9):1135-41. doi: 10.7205/MILMED-D-15-00518. PMID 27612365
- [Background] Miller JV, Andre Q, Timmers I, Simons L, Rasic N, Lebel C, Noel M. Subclinical post-traumatic stress symptomology and brain structure in youth with chronic headaches. Neuroimage Clin. 2021;30:102627. doi: 10.1016/j.nicl.2021.102627. Epub 2021 Mar 13. PMID 33812302
- [Background] Muldoon OT, Lowe RD, Jetten J, Cruwys T, Haslam SA. Personal and Political: Post-Traumatic Stress Through the Lens of Social Identity, Power, and Politics. Polit Psychol. 2021 Jun;42(3):501-533. doi: 10.1111/pops.12709. Epub 2020 Dec 13. PMID 34219849
- [Background] Mulvaney SW, Lynch JH, Hickey MJ, Rahman-Rawlins T, Schroeder M, Kane S, Lipov E. Stellate ganglion block used to treat symptoms associated with combat-related post-traumatic stress disorder: a case series of 166 patients. Mil Med. 2014 Oct;179(10):1133-40. doi: 10.7205/MILMED-D-14-00151. PMID 25269132
- [Background] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083
- [Background] Rauch SA, Eftekhari A, Ruzek JI. Review of exposure therapy: a gold standard for PTSD treatment. J Rehabil Res Dev. 2012;49(5):679-87. doi: 10.1682/jrrd.2011.08.0152. PMID 23015579
- [Background] Ross RJ, Ball WA, Dinges DF, Kribbs NB, Morrison AR, Silver SM, Mulvaney FD. Rapid eye movement sleep disturbance in posttraumatic stress disorder. Biol Psychiatry. 1994 Feb 1;35(3):195-202. doi: 10.1016/0006-3223(94)91152-5. PMID 8173020
- [Background] Ryff, C. D. (1989). Happiness is everything, or is it? Explorations on the meaning of psychological well-being. Journal of Personality and Social Psychology, 57(6), 1069.
- [Background] Schoenfeld FB, Marmar CR, Neylan TC. Current concepts in pharmacotherapy for posttraumatic stress disorder. Psychiatr Serv. 2004 May;55(5):519-31. doi: 10.1176/appi.ps.55.5.519. PMID 15128960
- [Background] Stein PK, Pu Y. Heart rate variability, sleep and sleep disorders. Sleep Med Rev. 2012 Feb;16(1):47-66. doi: 10.1016/j.smrv.2011.02.005. Epub 2011 Jun 11. PMID 21658979
- [Background] von der Warth R, Dams J, Grochtdreis T, Konig HH. Economic evaluations and cost analyses in posttraumatic stress disorder: a systematic review. Eur J Psychotraumatol. 2020 May 29;11(1):1753940. doi: 10.1080/20008198.2020.1753940. PMID 33488993
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 10(4).
- [Background] Williams DP, Koenig J, Carnevali L, Sgoifo A, Jarczok MN, Sternberg EM, Thayer JF. Heart rate variability and inflammation: A meta-analysis of human studies. Brain Behav Immun. 2019 Aug;80:219-226. doi: 10.1016/j.bbi.2019.03.009. Epub 2019 Mar 11. PMID 30872091